CLINICAL TRIAL: NCT06210087
Title: The Effect of the Open-glottis (Spontaneous) Pushing Technique Versus the Closed-glottis (Valsalva) Pushing Technique in the Second Stage of Labor on Fetal Acid-base Level and Maternal Outcomes: a Randomized Controlled Trial
Brief Title: Open-glottis Pushing Technique Versus the Valsalva Pushing Technique in the Second Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ayla Kanbur, Principal Investigator (Assoc. Dr.), Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: VALSPONPUSH
Record Dates: First submitted 2023-12-22; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Evidence-Based Practice; Labor; Prolonged, Second Stage; Labor; Fetal Acidosis Complicating Labor and Delivery

STUDY DESIGN:
Intervention Model Description: Spontaneous pushing-Experimental Group Valsalva-type pushing-Control Group
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spontaneous pushing (Experimental): The researcher provided training on the spontaneous pushing technique to the pregnant women selected for the experimental group in the first stage of labor and showed how to do it. During the second stage of labor, the women were encouraged and supported in this direction.
  Interventions: Other: Spontaneous pushing technique
- Valsalva-type pushing (No Intervention): Routine procedures of the delivery room were performed on the pregnant women in the control group, and the researcher carried out no intervention.

INTERVENTIONS:
Other: Spontaneous pushing technique — Pregnant women selected for the experimental group were trained on spontaneous pushing technique in the first stage of labor. During the second stage of labor, the women were encouraged and supported in this direction.
  Arms: Spontaneous pushing

SUMMARY:
Pushing has been discussed for decades, primarily in terms of facilitating care in the second stage of labor and maternal/fetal outcomes.

Valsalva-type pushing is the pushing performed by a pregnant woman by holding her breath. Various physiological findings argue against the Valsalva maneuver may adversely affect the acid-base balance and cerebral oxygenation of the fetus. It has been shown that a long apnea period (long closed glottis) associated with the Valsalva maneuver during the expulsive stage of labor increases lactate concentration in the mother and the fetus and adversely affects the fetal acid-base balance.

Spontaneous pushing is the pushing movements that occur naturally in the second stage of birth. Spontaneous pushing is part of the natural birth process and encourages women to trust the natural functioning of their bodies. When pushing with an open glottis, fetal placental circulation is preserved since the pressure on the chest does not increase and there are fewer hemodynamic effects.

The World Health Organization (WHO) recommends that women in the second stage of labor should be encouraged and supported to follow their pushing urges. The WHO states that healthcare professionals involved in obstetric care should avoid the Valsalva maneuver due to the lack of evidence that this technique has any benefit in the second stage of labor. The WHO supports spontaneous pushing in its recommendations for a positive birth experience. Safe termination of labor for both the mother and fetus is one of the primary duties of all healthcare professionals. There are few studies examining the maternal and fetal effects of the pushing types used during labor, especially their effects on the acid-base balance in the fetus. To contribute to the quality of evidence on the subject, the effects of Valsalva-type and spontaneous pushing techniques in the second stage of labor on fetal acid-base level and maternal outcomes were examined.

Hypotheses of the Research H1: Spontaneous pushing reduces the mother's pain level. H2: Spontaneous pushing increases the mother's birth satisfaction. H3: Spontaneous pushing positively affects the acid-base balance of the fetus. H4: Valsalva-type pushing increases the mother's pain level. H5: Valsalva-type pushing reduces the mother's birth satisfaction. H6: Valsalva-type pushing negatively affects the acid-base balance of the fetus.

ELIGIBILITY:
Inclusion Criteria:

Being at least a primary school graduate, being between the 38th and 42nd weeks of gestation, having a single fetus in a vertex position, giving vaginal birth, not developing any complications during labor, and volunteering to participate in the study.

Exclusion Criteria:

High-risk pregnancy, developing complications during labor, and having a diagnosed psychiatric disease.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 162 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | During the data collection period of 7 months
  for labor pain level
  Visual Analogue Scale (VAS): It is used to measure the intensity of pain in the patient. The VAS is a measurement tool that is frequently and safely used to evaluate labor pain. The VAS is 10 cm long. Women were asked to score pain from zero to 10. A zero score means no pain, while 10 means the most severe pain experienced.
  Pain level was evaluated with the VAS in the 2nd Stage of Labor.
questionnaire-Postpartum Interview Form | During the data collection period of 7 months
  for mother's birth satisfaction
  Postpartum Interview Form: It is a form consisting of questions that include women's opinions about the pushing type applied during labor.
  The postpartum interview form was applied to women in the experimental and control groups during the fourth stage of labor.
blood samples-Examination of blood samples in the laboratory | During the data collection period of 7 months
  acid-base balance of the fetus
  In the experimental and control groups, after the umbilical cord was clamped in the third stage of birth, 1 cc blood samples were taken from the umbilical blood.
  Blood samples for fetal acid base measurement were taken in the 3rd stage of labor.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla Kanbur, PhD, Study Director — Ataturk University; Özlem Koç, PhD, Principal Investigator — Tarsus University; Sibel EJDER TEKGÜNDÜZ, Dr., Study Chair — University of Health Science, Faculty of Medicine, Erzurum City Hospital; Özlem Selime MERTER, PhD, Study Chair — Firat University; Serap EJDER APAY, Study Director — Ataturk University
Locations (1):
- Fırat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
individual participant data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication